CLINICAL TRIAL: NCT03988296
Title: Adapting Novel Molecular Diagnostic Methods for Detection of Plasmodium Knowlesi in Sarawak, Malaysia
Brief Title: Molecular Diagnostic Methods for Detection of Plasmodium Knowlesi
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00102072
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-06

CONDITIONS: Plasmodium Knowlesi Infection
Keywords: Monkey malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 5ml Whole blood samples will be collected in a labeled EDTA acid tube. A minimum of 250ul of whole blood will be used to prepare dried blood spots on filter cards at the time of patient enrollment in the respective hospital. Extracted DNA from the remaining whole blood sample will be used to conduct molecular assays at Clinical Research Centre Sibu Hospital. Extracted DNA will be tested with the new single-step polymerase chain reaction (PCR) and the nested PCR at Sibu Hospital. An aliquot of same DNA will be shipped on dry ice to the CDC (Georgia, USA) for performing photo-induced electron transfer - polymerase chain reaction (PET-PCR) assays
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the sensitivity, specificity, and practical value of two new molecular diagnostic assays compared to a more classical nested molecular diagnostic assay and the routine microscopy (both of which are the current gold standard) in detection of P. knowlesi.

ELIGIBILITY:
Inclusion Criteria:

* Suspected for malaria infection; fever (axillary or tympanic temperature ≥ 37.5 °C or oral or rectal temperature of ≥ 38 °C) with chills, worsening malaise, headache lassitude, fatigue, abdominal discomfort, muscle and joint aches, anorexia, perspiration, or vomiting at the time of evaluation or within the past 48 hours
* Written informed consent is obtained.
* For Children (>7 to <18 years): parent or legal guardian provides written informed consent.

Exclusion Criteria:

* Patients living in, or returning from malaria endemic area outside of Sarawak within 2 weeks of illness onset
* They have a clear alternative diagnosis other than malaria by a trained health care professional.

Min Age: 7 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Both adults and children > 7 years old suspected for malaria and meeting inclusion criteria will be eligible to participate. Study subjects will be enrolled at Sarawak Hospitals, both hospitalized and outpatients, using an informed consent process (or assent for children 7-18 years) that permits the completion of a brief questionnaire and collection of a blood sample.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Number of patients with a possible diagnosis of malaria | 10 weeks
  Possible diagnosis of malaria as defined in accordance with the inclusion and exclusion criteria. Giemsa-stained thick and thin smears will be prepared for verification of parasitaemia by microscopy in the respective hospital laboratories

SECONDARY OUTCOMES:
Statistical association between risk factors and diagnostic assays results. | 10 weeks
  A brief enrollment questionnaire will be used to determine a statistical association between demographic and behavioral/occupational risk factors and the assays results combined

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C. Gray, MD, Principal Investigator — Duke University Medical Centre
Locations (3):
- Malaysia (3):
  - Kapit Hospital, Kapit, Sarawak
  - Sarikei Hospital, Sarikei, Sarawak
  - Sibu Hospital, Sibu, Sarawak

IPD SHARING:
Plan to Share IPD: No
Subjects' anonymity will be maintained and confidentiality of records and documents that could identify subjects will be protected, respecting the privacy and confidentiality rules in accordance with applicable regulatory requirements. Only the site principle investigators will be able to backlink the study data to the patient's medical record.

REFERENCES:
- [Background] Richards J, Mueller I. Identifying the risks for human transmission of Plasmodium knowlesi. Lancet Planet Health. 2017 Jun;1(3):e83-e85. doi: 10.1016/S2542-5196(17)30053-0. Epub 2017 Jun 9. No abstract available. PMID 29851611
- [Background] Imai N, White MT, Ghani AC, Drakeley CJ. Transmission and control of Plasmodium knowlesi: a mathematical modelling study. PLoS Negl Trop Dis. 2014 Jul 24;8(7):e2978. doi: 10.1371/journal.pntd.0002978. eCollection 2014 Jul. PMID 25058400
- [Background] Singh B, Daneshvar C. Human infections and detection of Plasmodium knowlesi. Clin Microbiol Rev. 2013 Apr;26(2):165-84. doi: 10.1128/CMR.00079-12. PMID 23554413
- [Background] Singh B, Kim Sung L, Matusop A, Radhakrishnan A, Shamsul SS, Cox-Singh J, Thomas A, Conway DJ. A large focus of naturally acquired Plasmodium knowlesi infections in human beings. Lancet. 2004 Mar 27;363(9414):1017-24. doi: 10.1016/S0140-6736(04)15836-4. PMID 15051281
- [Background] Barber BE, William T, Grigg MJ, Yeo TW, Anstey NM. Limitations of microscopy to differentiate Plasmodium species in a region co-endemic for Plasmodium falciparum, Plasmodium vivax and Plasmodium knowlesi. Malar J. 2013 Jan 8;12:8. doi: 10.1186/1475-2875-12-8. PMID 23294844
- [Background] Komaki-Yasuda K, Vincent JP, Nakatsu M, Kato Y, Ohmagari N, Kano S. A novel PCR-based system for the detection of four species of human malaria parasites and Plasmodium knowlesi. PLoS One. 2018 Jan 25;13(1):e0191886. doi: 10.1371/journal.pone.0191886. eCollection 2018. PMID 29370297
- [Background] Lucchi NW, Poorak M, Oberstaller J, DeBarry J, Srinivasamoorthy G, Goldman I, Xayavong M, da Silva AJ, Peterson DS, Barnwell JW, Kissinger J, Udhayakumar V. A new single-step PCR assay for the detection of the zoonotic malaria parasite Plasmodium knowlesi. PLoS One. 2012;7(2):e31848. doi: 10.1371/journal.pone.0031848. Epub 2012 Feb 20. PMID 22363751
- [Background] Lucchi NW, Narayanan J, Karell MA, Xayavong M, Kariuki S, DaSilva AJ, Hill V, Udhayakumar V. Molecular diagnosis of malaria by photo-induced electron transfer fluorogenic primers: PET-PCR. PLoS One. 2013;8(2):e56677. doi: 10.1371/journal.pone.0056677. Epub 2013 Feb 20. PMID 23437209